CLINICAL TRIAL: NCT01116284
Title: Laparoscopic Suture Plication of an Enlarged Gastric Stoma in the Gastric Bypass Patient
Brief Title: Laparoscopic Revision of an Enlarged Gastric Outlet After Gastric Bypass
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no patients to recruit
Sponsor: Baystate Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BH-10-016
Record Dates: First submitted 2010-05-03; First posted 2010-05-04 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Morbid Obesity
Keywords: Weight Loss; Obesity; Gastric Bypass
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Revision of gastric bypass (Experimental): A laparoscopic plication of the gastrojejunostomy will be performed after three 5-mm trocars are placed in the upper abdomen. Then using Ethibond suture, laparoscopic plication of the gastrojejunostomy on the medial, lateral and anterior surface of the anastomosis will be performed. The resulting anastomosis will be evaluated with intraoperative endoscopy and leak tested intraoperatively. The patients will be evaluated in the post-operative period with an expected discharge from the hospital within 24 hours.
  Interventions: Procedure: Revision of gastric bypass

INTERVENTIONS:
Procedure: Revision of gastric bypass — A laparoscopic operation will be performed to decrease the size of the enlarged gastric outlet. Three 5-mm laparoscopic trocars will be placed in the upper abdomen and suture plication of the gastrojejunostomy on the medial, lateral and anterior surface of the anastomosis will be performed. The resulting anastomosis will be evaluated with intraoperative endoscopy and leak tested intraoperatively. The patients will be evaluated in the post-operative period and are expected to be discharged from the hospital within 24 hours.
  Other Names: Laparoscopic plication of gastrojejunostomy

SUMMARY:
The purpose of this study is to determine if laparoscopic plication of a gastrojejunostomy is an effective surgical option for the Roux-en-Y gastric bypass patient who has regained weight due to a dilated gastric stoma. There are several reasons postulated to be the cause in patients who regain their weight after gastric bypass, including poor diet choices, dilation of the gastric pouch and enlargement of the gastric stoma. We aim to demonstrate that laparoscopic plication of the enlarge gastrojejunostomy can provide a safe and effective method to promote increased weight loss in this subset of gastric bypass patients.

DETAILED DESCRIPTION:
Excess body weight has been shown to have many adverse health effects including, increased risk of diabetes, hypertension, joint problems and early death. Roux-en-Y gastric bypass has been shown in the literature to be an effective weight loss surgery in the majority of patients who are morbidly obese in both short and long term weight loss management. However, while 80% of patients who undergo gastric bypass lose 67-75% of their excess body weight within 2 years of surgery, 20% of patients fail to loose or regain a substantial portion of their excess body weight.1-2 There are several reasons postulated to be the cause in patients who regain their weight after gastric bypass surgery. These include poor nutritional choices and eating high caloric carbohydrates in a grazing eating pattern. Also dilation of the gastric pouch overtime which can decrease the feeling of satiety and allow for larger meals to be eaten can cause recidivism of obesity. Another problem that can occur is the enlargement of the gastrojejunostomy anastomosis. Patients who have an opening larger than 2 cm can have rapid emptying of food into the intestines and decreased satiety with meals.

Plication is a standard surgical technique of folding or tucking in, which has been used widely on other parts of the human anatomy. There have been several methods tried in the past to place plication sutures in the gastrojejunostomy from an endoluminal approach.3-7 These devices have had some success but are not widely used at this time. We aim to demonstrate that laparoscopic suture plication of the enlarged gastrojejunostomy can provide a safe and effective minimally invasive method to promote increased weight loss in this subset of gastric bypass patients who have an enlarged gastric stoma.

Specific Aim 1 To demonstrate that the laparoscopic plication of an enlarged gastric bypass is a safe surgical option to promote weight loss in the Roux-en-Y gastric bypass patient.

Specific Aim 2 To monitor the effectiveness of long term weight loss after laparoscopic plication of the gastrojejunostomy in the Roux-en-Y gastric bypass patient

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patients 18 to 65 years old who are able to provide informed consent for this surgical procedure
2. Patients who have previously had a laparoscopic or open Roux-en-Y gastric bypass surgery
3. Patients who have regained or failed to lose their excess body weight

Exclusion Criteria:

1. Inability to provide informed consent
2. Patients who have dilated gastric pouch.
3. Patients who have a gastrogastric fistula.
4. Patients who are pregnant or plan to become pregnant during the follow up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Weight loss after revision of the gastric outlet | One Year
  To monitor the effectiveness of long term weight loss after laparoscopic plication of the gastrojejunostomy in the Roux-en-Y gastric bypass patient

SECONDARY OUTCOMES:
Safety of laparoscopic plication of a gastrojejunostomy | One year
  To demonstrate that the laparoscopic plication of an enlarged gastrojejunostomy is a safe surgical option to promote weight loss in the Roux-en-Y gastric bypass patient.

CONTACTS AND LOCATIONS:
Overall Officials: Burritt L Haag III, MD, Principal Investigator — Pioneer Valley Surgical Associates
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pioneer Valley Surgical Associates, P.C. — http://www.pvsurgical.com/
- See also: Baystate Medical Center — http://baystatehealth.com/Baystate